CLINICAL TRIAL: NCT02802046
Title: Evaluation of the Correlation Between the Coronary Stenosis Degree With FFRCT and the Grade of Stable Angina Pectoris
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guiyang No.4 People's Hospital (Other)
Responsible Party: Principal Investigator, Tan Song, Deputy director, Department of Radiology, Guiyang No.4 People's Hospital
Other Study IDs: 42925078-2
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Coronary Stenosis; Angina Pectoris
Keywords: FFRCT; Angina pectoris grade; Fractional flow reserve; CCTA
MeSH Terms: conditions — Coronary Stenosis; Angina Pectoris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FFR≦0.8: FFR is a score of 0 to 1, FFR < 0.75, has proved almost always accompanied by myocardial ischemia.
  Interventions: Radiation: Computed tomographic angiography of coronary artery
- FFR>0.8: FFR > 0.80 almost never associated with myocardial ischemia.
  Interventions: Radiation: Computed tomographic angiography of coronary artery

INTERVENTIONS:
Radiation: Computed tomographic angiography of coronary artery

SUMMARY:
Angina pectoris is the most common clinical manifestation of coronary heart disease（CHD）, which is the main feature of chest pain caused by transient myocardial ischemia. Chronic stable angina pectoris is the degree, frequency, nature and cause of angina pectoris in patients with no significant change in a few weeks. The disease incidence is complex, difficult to diagnosis and treatment, clinical should be combined with various inspection methods for diagnosis and differential diagnosis. Fractional flow reserve of computerized tomographic scanning (FFRCT ) allows computerized tomographic scanning（CT） to scan the determination of coronary blood flow and blood pressure in the heart at rest and hyperemia, but no need to additional check or drugs. This technique has been used for noninvasive fractional flow reserve (FFR) in the calculation, assuming normal artery, calculated by the ratio of the maximum blood flow and blood flow of coronary artery stenosis of an artery. Along with the development and progress of computational fluid dynamics, in the resting state by computed tomographic angiography of coronary artery(CCTA) image data based, simulation of coronary artery maximal hyperemia and according to the 3-dimensional model of the traditional method of reconstruction of coronary arterial tree and ventricular muscle structure, and in order to calculated coronary blood flow and pressure. FFRCT is a novel non-invasive examination method, using computed tomographic angiography of coronary artery image data can be calculated FFR, and preliminary study proved that it has a high degree of correlation with traumatic FFR. Therefore, this study aims to evaluate the correlation between the degree of coronary stenosis and the grading of angina pectoris by noninvasive means --FFRCT, in order to provide a new idea for the diagnosis and differential diagnosis of coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* After computed tomographic angiography of coronary artery (CCTA) for the diagnosis of coronary heart disease patients

Exclusion Criteria:

* First, the patients with hematological diseases, infectious disease, end-stage renal disease and malignant tumor and other diseases. Second, the patients with acute myocardial infarction. Last, the percutaneous coronary intervention(PCI) and coronary artery bypass grafting (GABG) after the operation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From 2015 to 2017 in our hospital for clinical diagnosis of coronary heart disease and computed tomographic angiography of coronary artery(CCTA) examination of patients.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
FFR Value | 1 years

SECONDARY OUTCOMES:
CCS Class | 1 years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor CA, Fonte TA, Min JK. Computational fluid dynamics applied to cardiac computed tomography for noninvasive quantification of fractional flow reserve: scientific basis. J Am Coll Cardiol. 2013 Jun 4;61(22):2233-41. doi: 10.1016/j.jacc.2012.11.083. Epub 2013 Apr 3. PMID 23562923
- [Background] Pijls NH, De Bruyne B, Peels K, Van Der Voort PH, Bonnier HJ, Bartunek J Koolen JJ, Koolen JJ. Measurement of fractional flow reserve to assess the functional severity of coronary-artery stenoses. N Engl J Med. 1996 Jun 27;334(26):1703-8. doi: 10.1056/NEJM199606273342604. PMID 8637515
- [Background] Legalery P, Schiele F, Seronde MF, Meneveau N, Wei H, Didier K, Blonde MC, Caulfield F, Bassand JP. One-year outcome of patients submitted to routine fractional flow reserve assessment to determine the need for angioplasty. Eur Heart J. 2005 Dec;26(24):2623-9. doi: 10.1093/eurheartj/ehi484. Epub 2005 Sep 1. PMID 16141256